CLINICAL TRIAL: NCT00767728
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Trial to Evaluate the Use of Mesalamine Pellet Formulation 1.5G QD to Maintain Remission From Mild to Moderate Ulcerative Colitis
Brief Title: Mesalamine Pellet to Maintain Remission of Mild to Moderate Ulcerative Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Audrey Shaw, Ph.D., Salix Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MPUC3004
Record Dates: First submitted 2008-09-17; First posted 2008-10-07 (Estimated); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Ulcerative Colitis
Keywords: UC; ulcerative colitis; IBD; Inflammatory Bowel Disease
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Mesalamine pellets
  Interventions: Drug: Granulated mesalamine
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Granulated mesalamine — 0.375 g of mesalamine granules were encapsulated in a hard gelatin shell. 1.5 g of eMG (4 capsules) were administered orally QD, in the morning.
  Arms: 1
Drug: Placebo — Matching placebo capsules (4 capsules) were administered orally QD, in the morning.
  Arms: 2

SUMMARY:
The purpose of this study is to compare the maintenance of mild to moderate ulcerative colitis remission with six months of treatment with 1.5 grams of mesalamine pellets each day versus placebo.

DETAILED DESCRIPTION:
This is a Phase 3 study evaluating the effectiveness and safety of eMG 1.5 g given once daily (QD) compared to placebo in subjects with demonstrated remission from UC. Eligible subjects are randomized in a 2:1 ratio (active:placebo) to receive 1 or 2 treatments: 1.5g eMG (4 capsules total) or matching placebo capsules QD for 6 months.

The study consists of a screening phase (completed within 7 days prior to randomization), a treatment phase (6 months), and a follow-up visit (2 weeks after end-of-study [EOS] visit.) The treatment phase consists of 4 scheduled study visits: visit 1 (baseline/randomization (day 1), visit 2 (month 1), visit 3 (month 3), visit 4 (EOS (month 6).

Primary objective:

To compare the maintenance of remission from mild to moderate ulcerative colitis as measured by rectal bleeding and endoscopic mucosal appearance after 6 months of treatment with encapsulated mesalamine granules (eMG) of 1.5 g QD, as compared with placebo.

Secondary objective:

To compare the safety and tolerability of long-term dosing with eMG at 1.5 g QD as compared to placebo in the maintenance of remission from mild to moderate UC.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of ulcerative colitis and in remission for at least 1 month
* Greater than 18 years of age

Exclusion Criteria:

* Allergy/intolerance to aspirin, mesalamine, or other salicylates
* Prior bowel surgery other than appendectomy
* Pregnancy, at risk of pregnancy, or lactating
* HIV or hepatitis B or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2004-12; Primary Completion 2007-08 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Proportion of subject who were relapse free after 6 months of treatment | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Mexico, Missouri, United States

REFERENCES:
- [Derived] Zakko SF, Gordon GL, Murthy U, Sedghi S, Pruitt R, Barrett AC, Bortey E, Paterson C, Forbes WP, Lichtenstein GR. Once-daily mesalamine granules for maintaining remission of ulcerative colitis: pooled analysis of efficacy, safety, and prognostic factors. Postgrad Med. 2016;128(3):273-81. doi: 10.1080/00325481.2016.1152876. Epub 2016 Mar 1. PMID 26861051
- [Derived] Lichtenstein GR, Gordon GL, Zakko S, Murthy U, Sedghi S, Pruitt R, Barrett AC, Bortey E, Paterson C, Forbes WP. Long-Term Benefit of Mesalamine Granules for Patients Who Achieved Corticosteroid-Induced Ulcerative Colitis Remission. Dig Dis Sci. 2016 Jan;61(1):221-9. doi: 10.1007/s10620-015-3866-7. Epub 2015 Nov 12. PMID 26563167
- [Derived] Lichtenstein GR, Zakko S, Gordon GL, Murthy U, Sedghi S, Pruitt R, Merchant K, Bortey E, Forbes WP. Mesalazine granules 1.5 g once-daily maintain remission in patients with ulcerative colitis who switch from other 5-ASA formulations: a pooled analysis from two randomised controlled trials. Aliment Pharmacol Ther. 2012 Jul;36(2):126-34. doi: 10.1111/j.1365-2036.2012.05142.x. Epub 2012 May 23. PMID 22617015